CLINICAL TRIAL: NCT06987760
Title: Comparing Different Diameter fURSs With Similar RESDs for the Treatment of Upper Urinary Tract Stones - A Randomized Controlled Multi-center Clinical Trials
Brief Title: Comparing Different Diameter fURSs With Similar RESDs for the Treatment of Upper Urinary Tract Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: The First People's Hospital of Fuyang District, Hangzhou City (Unknown); The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MNWK202401
Record Dates: First submitted 2025-02-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-02

CONDITIONS: Ureter Injury; Urolithiasis; Lower Urinary Tract; Efficacy, Self
Keywords: Urolithiasis; Ratio of Endoscope-Sheath Diameter; Flexible ureteroscope
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: 7.5Fr disposable electronic flexible ureteroscope combine with 10Fr distally deflectable ureteral access sheath.
Who Masked: Participant
Masking Description: 9.0Fr disposable electronic flexible ureteroscope combine with 12Fr distally deflectable ureteral access sheath.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 7.5Fr fURS and 10Fr UAS (Experimental): 7.5Fr disposable electronic flexible ureteroscope combine with 10Fr distally deflectable ureteral access sheath.
  Interventions: Procedure: flexible ureteroscope urolithiasis
- 9.0Fr fURS and 12Fr UAS (Active Comparator): 9.0Fr disposable electronic flexible ureteroscope combine with 12Fr distally deflectable ureteral access sheath.
  Interventions: Procedure: flexible ureteroscope urolithiasis

INTERVENTIONS:
Procedure: flexible ureteroscope urolithiasis — Using flexible ureteroscope combine with urethral access sheath to treatment urolithiasis

SUMMARY:
Comparing the Efficiency, Effectiveness, and Safety of fURS lithotripsy with Similar RESDs in the Treatment of Upper Urinary Tract Stones.

DETAILED DESCRIPTION:
Comparing the Efficiency, Effectiveness, and Safety of fURS lithotripsy with Similar RESDs in the Treatment of Upper Urinary Tract Stones.

ELIGIBILITY:
Inclusion Criteria:

- 1.Patients with kidney stones or upper ureteral stones with a cumulative diameter of less than 3 cm are selected for ureteral soft lens holmium laser lithotripsy.

2.Age 18 to 80 years old, gender unlimited. 3.The subjects have no mental illness or language dysfunction, can understand the situation of the study and can sign informed consent.

Exclusion Criteria:

* 1.Patients with a history of ureteral stenosis or who have undergone open or laparoscopic ureteral or renal lithotomy.

  2.Patients with fever one week before surgery 3.Pregnant women and menstruating patients. 4.Patients with combined systemic disease or inability to tolerate anesthesia. 5.Patients undergoing simultaneous surgery for bilateral upper urinary tract stones.

  6.Patients with ureteral stent indwelling before surgery. 7.In patients with severe hydronephrosis, the separation of the renal collecting system is greater than 4 cm.

  8.Patients with renal anatomic malformations such as polycystic kidney, horseshoe kidney, and ectopic kidney.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of ureteral access sheath insertion | From enrollment to completion of surgery
  Proportion of successful ureteral implantation, success rate = number of successful cases/total number of cases

SECONDARY OUTCOMES:
The condition of ureter injury | 24 hours
  The ureter was observed at exit of the ureteroscope and graded according to Traxer's proposed grading system.
Stone clearance rate | up to 8 weeks.
  Residual stones less than 4 mm are considered to be free of residual stones.
Operation time | 24 hours
  The duration of the operation from start to finish.
The incidence of surgical complications | 7 days
  The occurrence of postoperative fever, urogenic sepsis and septic shock

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China